CLINICAL TRIAL: NCT00143962
Title: Comparison of Two Approaches to Weight Loss Follow-Up Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 801787; NCT00200811 (obsolete NCT alias)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Obesity
Keywords: Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Diet, Carbohydrate-Restricted

INTERVENTIONS:
Behavioral: Low Carbohydrate Diet

SUMMARY:
This is a follow-up research study to determine if there are any differences in the long-term maintenance of two diet groups, the Atkins' diet (low-carbohydrate) or the LEARN program (low-fat). The Atkins' diet continues to get a significant amount of popular attention and very little scientific evaluation. Due to the small amount of scientific data to support a low-carbohydrate diet and given the wide spread use of this type of diet, it is important to evaluate the long-term safety and effectiveness of the Atkins' diet.

We will evaluate whether there are any differences between these two groups 3-years after participation in the initial 1-year study period. We will specifically assess weight, cholesterol levels, glucose and insulin levels, and eating habits and mood as we did originally.

DETAILED DESCRIPTION:
***PLEASE NOTE: Only those who participated in the original study of low carbohydrate and low fat diets are eligable for enrollment in this follow-up study***

ELIGIBILITY:
Inclusion Criteria

* Body mass index between 30 and 40
* Live and work within 1 hour of the study site
* Stable psychological status Exclusion criteria
* History of heart disease, heart attack, or stroke
* Blood pressure >140/90 mmHg
* Abnormal cholesterol levels
* Significant psychiatric illness
* Any medication that affects weight or metabolic rate
* Presence or history of a chronic disease that is known to affect appetite, food intake, or metabolism (i.e., diabetes, thyroid disease, or cancer)
* Currently using antidepressants, steroids, tobacco, or illegal drugs
* Pregnant, breastfeeding, or planning pregnancy
* 10 lb change in weight within 6 months of study entry
* History of malignant arrhythmias or cerebrovascular, renal, or hepatic disease
* History of protein wasting diseases or gout
* Severe arthritis
* Osteoporosis
* Certain types of hormone replacement therapy
* Currently following a vegetarian diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-07; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Obesity

CONTACTS AND LOCATIONS:
Overall Officials: Gary Foster, PhD, Principal Investigator — University of Pennsylvania; Holly Wyatt, MD, Principal Investigator — University of Colorado, Denver; James Hill, PhD, Principal Investigator — University of Colorado, Denver; Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - University of Colorado, Denver, Colorado
  - Washington University, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Foster GD, Wyatt HR, Hill JO, McGuckin BG, Brill C, Mohammed BS, Szapary PO, Rader DJ, Edman JS, Klein S. A randomized trial of a low-carbohydrate diet for obesity. N Engl J Med. 2003 May 22;348(21):2082-90. doi: 10.1056/NEJMoa022207. PMID 12761365